CLINICAL TRIAL: NCT04883918
Title: Evaluation of Safety and Efficacy of ASC930 in Patients With Steroid-Refractory Acute Graft Versus Host Disease
Brief Title: ASC930 in Patients With Steroid-Refractory Acute Graft Versus Host Disease (SR-aGVHD)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ASC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASC-aGVHD-001
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-01

CONDITIONS: Acute-graft-versus-host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ASC930 (Experimental): Experimental Arm
  Interventions: Biological: ASC930

INTERVENTIONS:
Biological: ASC930 — 4 intravenous doses of ASC930

SUMMARY:
Acute GVHD following allogeneic HCT is an immune-triggered process, leading to profound immune dysregulation and organ dysfunction. Despite pivotal advances, aGVHD is one of the leading causes of non-relapse mortality in patients undergoing HCT.

Placenta-derived DSCs, isolated from the fetal membrane of maternal origin, are a type of stromal cells with well-characterized immunosuppressive properties. The current study is designed to assess the safety and efficacy of 4 intravenous (IV) doses of ASC930 DSC cells in aGVHD patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥ 2 months of age
* Diagnosis of aGVHD grade II-IV following allogeneic HSCT according to standard criteria (Harris, 2016).
* Diagnosis of SR-aGVHD according to Mohty (2020)
* Meet one of the following criteria:

  * Participants who are Ruxolitinib-refractory, according to Mohty (2020)
  * Participants who are not eligible for SOC therapy
  * Participants who agree to receive ASC930 as a second-line therapy
* Karnofsky/Lansky Performance Status of at least 30 at the time of study entry
* Minor participants must be capable of giving written assent as appropriate per the applicable age (per local regulatory requirements).

Exclusion Criteria:

* Diagnosis of active Hepatic Sinusoidal Obstruction Syndrome (SOS)
* Presence of an active uncontrolled infection
* Active treatment for a hyprecoagulation disorder
* Evidence of diffuse alveolar hemorrhage or other active pulmonary disease
* Evidence of encephalopathy as defined by a change in mental status since the onset of aGVHD
* Evidence of relapse of malignancy
* Receival of agents other than steroids for primary treatment of aGVHD
* Severe allergic history to cell-based products

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) at Day 28 | 28 days post-infusion
Number of adverse events, and serious AEs | 30 days post-infusion

SECONDARY OUTCOMES:
Duration of response (DOR) at DAY 180 | 180 days post-infusion
Overall survival (OS) rate at DAY 180 | 180 days post-infusion
Complete Response (CR) at Day 28 and Day 180 | 28 and 180 days post-infusion

IPD SHARING:
Plan to Share IPD: No